CLINICAL TRIAL: NCT07319091
Title: Evaluation of Mitochondrial Metabolism in Patients With Cystinosis: CYSTI-MITO Project
Brief Title: Cystinosis and Mitochondrial Metabolism
Acronym: CYSTI-MITO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL25_0542
Record Dates: First submitted 2025-11-18; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Cystinosis; Native Kidney
Keywords: Cystinosis; Mitochondria; Cystinosis Metabolic Bone Disease (CMBD); Myopathy
MeSH Terms: conditions — Cystinosis; Muscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cystinosis patient (Other): Patient with genetically confirmed nephropathic cystinosis Men and women, children and adults with cystinosis Undergoing conservative treatment on native kidneys Age ≥ 2 years Patients receiving oral cysteamine Patients with social security coverage Informed consent signed by the participant or parents or legal guardians before participating in the study
  Interventions: Other: Mitochondrial metabolism

INTERVENTIONS:
Other: Mitochondrial metabolism — Study of membrane potential by flow cytometry of circulating monocyte cells and evaluate the respiratory chain of these cells in patients with cystinosis and described musculoskeletal disorders in the study population in clinical and biological terms including metabolomic analysis of patients' blood and urine

SUMMARY:
Cystinosis is a monogenic autosomal recessive lysosomal storage disease with complete penetrance, caused by a biallelic mutation in the CTNS gene (17p13.2) encoding cystinosin, a ubiquitous membrane protein whose role is to clear cystine into the cytosol. Its dysfunction in patients with cystinosis leads to systemic accumulation of cystine, an oxidised dimer of cysteines linked by a disulphide bridge, in the lysosomal space, and irreversible cellular dysfunction. Renal damage is at the forefront, with Fanconi syndrome (proximal tubulopathy) and chronic renal failure developing early in childhood/adolescence. There are also multi-systemic disorders, notably endocrine and ophthalmological. Cysteamine is an amino thiol which reduces the level of intra-lysosomal cystine by breaking the disulphide strands of cystine, giving two cysteines which complex with cysteamine to leave the lysosome. Since the late 1980s, there has been an immediate-release form of the drug, which has considerably improved overall patient survival despite having a major impact on quality of life. This improvement in survival has also led to the emergence of later complications that were not previously observed. This musculoskeletal complication (described in an international consensus in 2019), known as 'CMBD' for Cystinosis Metabolic Bone Disease, may be explained at least in part by an intrinsic defect in the osteoblast and osteoclast that contribute to the human bone phenotype. This intrinsic bone defect appears to be responsible for premature ageing. In order to identify potential future therapeutic targets for CMBD, it is essential to gain a better understanding of the underlying pathophysiological mechanisms.

To better understand premature aging in extra-renal damage in cystinosis, it seems relevant to investigate energy metabolism dysfunction, particularly mitochondrial dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Patient with genetically confirmed nephropathic cystinosis
* Men and women, children and adults with cystinosis
* Undergoing conservative treatment on native kidneys
* Age ≥ 2 years
* Patients receiving oral cysteamine
* Patients with social security coverage
* Informed consent signed by the participant or parents or legal guardians before participating in the study

Exclusion Criteria:

* Patient not complying with study procedures
* Transplant or dialysis patient
* Patient on anticalcineurin
* Pregnant or breast-feeding woman
* Person deprived of liberty by a judicial or administrative decision
* Person not affiliated to a social security scheme or beneficiaries of a similar scheme

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Membrane potential of circulating monocyte cells | 24 months
  Mitochondrial metabolism was assessed by measuring the membrane potential by flow cytometry of circulating monocyte cells between subjects with and without cystinosis.

SECONDARY OUTCOMES:
Oxygen consumption rate (OCR) of circulating monocytic cells | 24 months
  The oxygen consumption rate (OCR) of circulating monocytic cells is measured by the Seahorse method. This method also measures the extracellular acidification rate (ECAR) of cells. The oxygen consumption rate (OCR) and the extracellular acidification rate (ECAR) are used to assess the respiratory chain of the cells, which will be compared between subjects with and without cystinosis.
Extracellular acidification rate (ECAR) of circulating monocytic cells | 24 months
  The extracellular acidification rate (ECAR) of circulating monocytic cells is measured by the Seahorse method. This method also measures the oxygen consumption rate (OCR) of cells. The extracellular acidification rate (ECAR) and the oxygen consumption rate (OCR) are used to assess the respiratory chain of the cells, which will be compared between subjects with and without cystinosis.
Age | 24 months
  The patient's age is a data used to produce a clinical description of musculoskeletal disorders based on current practice data such as : sex, weight, height, blood pressure, treatment, bone deformity, clinical sign of myopathy, grip strength test using the Grip-test (Z score) and the EAT10 (Eating Assessment Tool) questionnaire
Sex | 24 months
  The patient's sex is a data used to produce a clinical description of musculoskeletal disorders based on current practice data such as : age, weight, height, blood pressure, treatment, bone deformity, clinical sign of myopathy, grip strength test using the Grip-test (Z score) and the EAT10 (Eating Assessment Tool) questionnaire
Weight | 24 months
  The patient's weight is a data used to produce a clinical description of musculoskeletal disorders based on current practice data such as : age, sex, height, blood pressure, treatment, bone deformity, clinical sign of myopathy, grip strength test using the Grip-test (Z score) and the EAT10 (Eating Assessment Tool) questionnaire
Height | 24 months
  The patient's height is a data used to produce a clinical description of musculoskeletal disorders based on current practice data such as : age, sex, weight, blood pressure, treatment, bone deformity, clinical sign of myopathy, grip strength test using the Grip-test (Z score) and the EAT10 (Eating Assessment Tool) questionnaire
Blood pressure | 24 months
  The patient's blood pressure is a data used to produce a clinical description of musculoskeletal disorders based on current practice data such as : age, sex, weight, height, treatment, bone deformity, clinical sign of myopathy, grip strength test using the Grip-test (Z score) and the EAT10 (Eating Assessment Tool) questionnaire
Type of treatment | 24 months
  The patient's type of treatment is a data used to produce a clinical description of musculoskeletal disorders based on current practice data such as : age, sex, weight, height, blood pressure, bone deformity, clinical sign of myopathy, grip strength test using the Grip-test (Z score) and the EAT10 (Eating Assessment Tool) questionnaire
Bone deformity | 24 months
  The patient's bone deformity is a data used to produce a clinical description of musculoskeletal disorders based on current practice data such as : age, sex, weight, height, blood pressure, treatment, clinical sign of myopathy, grip strength test using the Grip-test (Z score) and the EAT10 (Eating Assessment Tool) questionnaire
Clinical sign of myopathy | 24 months
  Clinical sign of myopathy is a data used to produce a clinical description of musculoskeletal disorders based on current practice data such as : age, sex, weight, height, blood pressure, treatment, bone deformity, grip strength test using the Grip-test (Z score) and the EAT10 (Eating Assessment Tool) questionnaire
Grip-test score | 24 months
  The Grip-test is used to assess grip strength. Grip-test score is a data used to produce a clinical description of musculoskeletal disorders based on current practice data such as : age, sex, weight, height, blood pressure, treatment, bone deformity, clinical sign of myopathy and the EAT10 (Eating Assessment Tool) questionnaire
EAT10 (Eating Assessment Tool) questionnaire score | 24 months
  EAT10 (Eating Assessment Tool) questionnaire score is pathological if >= 3 :
  * 3-10 mild dysphagia
  * 11-20 moderate dysphagia
  * 21-40 severe dysphagia) questionnaire. EAT10 score is a data used to produce a clinical description of musculoskeletal disorders based on current practice data such as : age, sex, weight, height, blood pressure, treatment, bone deformity, clinical sign of myopathy and grip-test score
Complete ionogram | 24 months
  Complete ionogram is a data used to produce biological description of musculoskeletal disorders based on routine practice data such as C-reactive protein (CRP), intra-leukocyte cystine, Parathyroid hormone (PTH), total alkaline phosphatases, 25(OH) vitamin D, 1-25 (OH) vitamin D
C-Reactive Protein (CRP) | 24 months
  C-Reactive Protein (CRP) is a data used to produce biological description of musculoskeletal disorders based on routine practice data such as complete ionogram, intra-leukocyte cystine, Parathyroid hormone (PTH), total alkaline phosphatases, 25(OH) vitamin D, 1-25 (OH) vitamin D
Intra-leukocyte cystine | 24 months
  Intra-leukocyte cystine is a data used to produce biological description of musculoskeletal disorders based on routine practice data such as complete ionogram, C-Reactive Protein (CRP), Parathyroid hormone (PTH), total alkaline phosphatases, 25(OH) vitamin D, 1-25 (OH) vitamin D
Parathyroid hormone (PTH) | 24 months
  Parathyroid hormone (PTH) is a data used to produce biological description of musculoskeletal disorders based on routine practice data such as complete ionogram, C-Reactive Protein (CRP),intra-leukocyte cystine, total alkaline phosphatases, 25(OH) vitamin D, 1-25 (OH) vitamin D
Total alkaline phosphatases | 24 months
  Total alkaline phosphatases is a data used to produce biological description of musculoskeletal disorders based on routine practice data such as complete ionogram, C-Reactive Protein (CRP), intra-leukocyte cystine, Parathyroid hormone (PTH), 25(OH) vitamin D, 1-25 (OH) vitamin D
25(OH) vitamin D | 24 months
  25(OH) vitamin D is a data used to produce biological description of musculoskeletal disorders based on routine practice data such as complete ionogram, C-Reactive Protein (CRP), intra-leukocyte cystine, Parathyroid hormone (PTH), total alkaline phosphatases, 1-25 (OH) vitamin D
1-25 (OH) vitamin D | 24 months
  1-25 (OH) vitamin D is a data used to produce biological description of musculoskeletal disorders based on routine practice data such as complete ionogram, C-Reactive Protein (CRP), intra-leukocyte cystine, Parathyroid hormone (PTH), total alkaline phosphatases, 25 (OH) vitamin D
Distribution of plasma organic amino acids | 24 months
  Study of metabolomic analysis of patients' blood
Distribution of urinary organic amino acids | 24 months
  Study of metabolomic analysis of patients' urine
Urinary Krebs cycle intermediate metabolites | 24 months
  Study of metabolomic analysis of patients' urine

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Service de néphrologie pédiatrique, Hôpital Femme Mère Enfant, Hospices Civils de Lyon, Bron
  - Service de Néphrologie pédiatrique, Hôpital Jeanne de Flandre, Lille
  - Service de néphrologie et exploration fonctionnelle rénale, Hôpital Edouard Herriot, Hospices Civils de Lyon, Lyon
  - Service de Néphrologie pédiatrique, Hôpital de la Timone, Marseille
  - Service de Néphologie et endocrinologie pédiatrique, Hôpital Arnaud de Villeneuve, Montpellier
  - Service de Néphrologie pédiatrique, Hôpital Necker-Enfants Malades, Paris
  - Service de Néphrologie-transplantation rénale adultes, Hôpital Necker-Enfants Malades, Paris
  - Service de Néphrologie pédiatrique, Hôpital Robert Debré, Paris
  - Service de Néphrologie-Dialyse-Transplantation pédiatrique, Hôpital d'enfants Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No